CLINICAL TRIAL: NCT02115516
Title: Safety and Protective Efficacy of Intravenous Immunization With Cryopreserved Plasmodium Falciparum Sporozoites Under Chemoprophylaxis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Institute of Tropical Medicine, University of Tuebingen (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TUCHMI-002; 2013-003900-38 (EudraCT Number)
Record Dates: First submitted 2014-04-11; First posted 2014-04-16 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2016-02

CONDITIONS: Malaria; Plasmodium Falciparum Malaria
Keywords: Malaria; Plasmodium falciparum malaria; Antimalarial chemoprophylaxis; PfSPZ Challenge; Cryopreserved Plasmodium Falciparum Sporozoites; PfSPZ-CVac
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Stage A: Grp A1 - 3,200 PfSPZ Challenge (Experimental): Group A1 (PfSPZ Challenge) (n=9) receives three injections of 3,200 PfSPZ Challenge intravenous (IV) at 4-week intervals. Immunizations are given under a standard chemoprophylactic regimen with chloroquine. Two days before the first PfSPZ Challenge injection volunteers receive one oral dose of 10 mg/kg CQ base. On Day 5 volunteers will receive 5 mg/kg CQ base. Subsequently, volunteers will receive 5 mg/kg CQ base in weekly intervals for a total of ten doses. Eight weeks after the last immunization, volunteers will undergo homologous CHMI with 3,200 PfSPZ Challenge IV. Early unblinding for this group may be done on Week 19, if required. All groups in Stage A are scheduled to be unblinded on Week 27.
  Interventions: Biological: PfSPZ Challenge
- Stage A: Grp A2 - 12,800 PfSPZ Challenge (Experimental): Group A2 (PfSPZ Challenge) (n=9) starts when Group A1 receives the second immunization. Group A2 receives three injections of 12,800 PfSPZ Challenge IV at 4-week intervals. Immunizations are given under a standard chemoprophylactic regimen with chloroquine. Two days before the first PfSPZ Challenge injection volunteers receive one oral dose of 10 mg/kg CQ base. On Day 5 volunteers will receive 5 mg/kg CQ base. Subsequently, volunteers will receive 5 mg/kg CQ base in weekly intervals for a total of ten doses. Eight weeks after the last immunization, volunteers will undergo homologous CHMI with 3,200 PfSPZ Challenge IV. Early unblinding for this group may be done on Week 23, if required. All groups in Stage A are scheduled to be unblinded on Week 27.
  Interventions: Biological: PfSPZ Challenge
- Stage A: Grp A3 - 51,200 PfSPZ Challenge (Experimental): Group A3 (PfSPZ Challenge) (n=9) starts when Group A2 receives the second immunization. Group A3 receives three injections of 51,200 PfSPZ Challenge IV at 4-week intervals. Immunizations are given under a standard chemoprophylactic regimen with chloroquine. Two days before the first PfSPZ Challenge injection volunteers receive one oral dose of 10 mg/kg CQ base. On Day 5 volunteers will receive 5 mg/kg CQ base. Subsequently, volunteers will receive 5 mg/kg CQ base in weekly intervals for a total of ten doses. Eight weeks after the last immunization, volunteers will undergo homologous CHMI with 3,200 PfSPZ Challenge IV. This group is scheduled to be unblinded with all other groups in Stage A Week on 27.
  Interventions: Biological: PfSPZ Challenge
- Stage A: Grp A1 - 0.9% Sodium Chloride (Placebo Comparator): Group A1 (placebo) (n=5) receives three injections of 0.9% Sodium chloride IV at 4 week intervals. Placebo injections are given under a standard chemoprophylactic regimen with chloroquine. Two days before the first placebo injection volunteers receive one oral dose of 10 mg/kg CQ base. On Day 5 volunteers will receive 5 mg/kg CQ base. Subsequently, volunteers will receive 5 mg/kg CQ base in weekly intervals for a total of ten doses. Eight weeks after the last placebo injection, volunteers will undergo homologous CHMI with 3,200 PfSPZ Challenge IV. Early unblinding for this group may be done on Week 19, if required. All groups in Stage A are scheduled to be unblinded on Week 27.
  Interventions: Biological: 0.9% Sodium Chloride (Placebo)
- Stage A: Grp A2 - 0.9% Sodium Chloride (Placebo Comparator): Group A2 (placebo) (n=5) starts when Group A1 receives the second immunization. Group A2 receives three injections of 0.9% Sodium chloride IV at 4 week intervals. Placebo injections are given under a standard chemoprophylactic regimen with chloroquine. Two days before the first placebo injection volunteers receive one oral dose of 10 mg/kg CQ base. On Day 5 volunteers will receive 5 mg/kg CQ base. Subsequently, volunteers will receive 5 mg/kg CQ base in weekly intervals for a total of ten doses. Eight weeks after the last placebo injection, volunteers will undergo homologous CHMI with 3,200 PfSPZ Challenge IV. Early unblinding for this group may be done on Week 23, if required. All groups in Stage A are scheduled to be unblinded on Week 27.
  Interventions: Biological: 0.9% Sodium Chloride (Placebo)
- Stage A: Grp A3 - 0.9% Sodium Chloride (Placebo Comparator): Group A3 (placebo) (n=5) starts when Group A2 receives the second immunization. Group A3 receives three injections of 0.9% Sodium chloride IV at 4 week intervals. Placebo injections are given under a standard chemoprophylactic regimen with chloroquine. Two days before the first placebo injection volunteers receive one oral dose of 10 mg/kg CQ base. On Day 5 volunteers will receive 5 mg/kg CQ base. Subsequently, volunteers will receive 5 mg/kg CQ base in weekly intervals for a total of ten doses. Eight weeks after the last placebo injection, volunteers will undergo homologous CHMI with 3,200 PfSPZ Challenge IV. This group is scheduled to be unblinded with all other groups in Stage A on Week 27.
  Interventions: Biological: 0.9% Sodium Chloride (Placebo)
- Stage B: Grp B1 - 51,200 PfSPZ Challenge (Experimental): Group B1 (n=5) will receive the optimal PfSPZ Challenge immunizing dose from the dose-escalation phase (Stage A; 51,200 PfSPZ Challenge (NF54)), using the same standard chemoprophylactic regimen with CQ (10 mg/kg CQ base loading dose, followed by weekly dosing with 5 mg/kg CQ base), but for five instead of ten weeks. Group B1 will receive 3 injections of 51,200 PfSPZ Challenge (NF54) on days 0, 14 and 28. All volunteers in Group B1 will undergo homologous CHMI with PfSPZ Challenge 10 weeks after the last immunization.
  Interventions: Biological: PfSPZ Challenge
- Stage B: Group B1 - 0.9% Sodium Chloride (Placebo Comparator): Group B1 (placebo) (n=2) will receive three injections of 0.9% Sodium Chloride on days 0, 14 and 28. This group will follow the the same standard chemoprophylactic regimen with CQ (10 mg/kg CQ base loading dose, followed by weekly dosing with 5 mg/kg CQ base), but for five instead of ten weeks. All volunteers in Group B1 will undergo homologous CHMI with PfSPZ Challenge 10 weeks after the last immunization.
  Interventions: Biological: 0.9% Sodium Chloride (Placebo)
- Stage B: Grp B2 - 51,200 PfSPZ Challenge (Experimental): Group B2 (n=5) will receive 3 injections of 51,200 PfSPZ Challenge on days 0, 14 and 28, using same std chemoprophylactic regimen with CQ (10 mg/kg CQ base loading dose, followed by weekly dosing with 5 mg/kg CQ base), for 5 instead of 10 wks. But Group B2 will receive extended-release azithromycin (ER-AZ, 2g) on the day of 1st PfSPZ Challenge and monitored for parasitemia by quantitative real time polymerase reaction (qPCR). In case that all CQ+ER-AZ treated volunteers are parasite-free until Day 11 following first PfSPZ Challenge injection, it will indicate that ER-AZ effectively killed the parasites in the liver prior to development of parasitemia. With demonstration of the effectiveness of ER-AZ, the 2nd and 3rd immunizations will be done under ER-AZ alone, otherwise CQ prophylaxis will continue and ER-AZ will not be administered for the 2nd and 3rd injections. Group B2 will undergo homologous CHMI with PfSPZ Challenge, 10 weeks after the last immunization.
  Interventions: Biological: PfSPZ Challenge
- Stage B: Group B2 - 0.9% Sodium Chloride (Placebo Comparator): Group B2 (placebo) (n=2) will receive three injections of 0.9% Sodium Chloride on days 0, 14 and 28, using the same standard chemoprophylactic regimen with CQ (10 mg/kg CQ base loading dose, followed by weekly dosing with 5 mg/kg CQ base), for 5 instead of 10 wks. But Group B2 will receive ER-AZ, 2g on the day of 1st placebo injection and monitored for parasitemia by qPCR. In case that all CQ+ER-AZ treated volunteers are parasite-free until Day 11 following 1st injection, it will indicate that ER-AZ effectively killed the parasites in the liver prior to the development of parasitemia. With demonstration of the effectiveness of ER-AZ, the 2nd and 3rd immunizations will be done under ER-AZ alone, otherwise CQ prophylaxis will be continued and ER-AZ will not be administered for 2nd and 3rd injections. Group B2 will undergo homologous CHMI with PfSPZ Challenge 10 weeks after last immunization.
  Interventions: Biological: 0.9% Sodium Chloride (Placebo)
- Stage B: Grp B3 - 51,200 PfSPZ Challenge (Experimental): Group B3 (n=9) volunteers will receive CQ and PfSPZ Challenge simultaneously every five days with one additional dose of CQ five days after the third PfSPZ Challenge injection. A 10 mg/kg CQ base loading dose is given at the time of first PfSPZ Challenge inoculation, followed by 5 mg/kg CQ base on the day of second and third inoculation and five days after the last PfSPZ Challenge inoculation. Group B3 will undergo homologous CHMI with PfSPZ Challenge 10 weeks after the last immunization.
  Interventions: Biological: PfSPZ Challenge
- Stage B: Group B3 - 0.9% Sodium Chloride (Placebo Comparator): Group B3 (placebo) (n=2) volunteers will receive CQ and 0.9% Sodium Chloride simultaneously every five days with one additional dose of CQ five days after the third placebo injection. A 10 mg/kg CQ base loading dose is given at the time of first placebo injection, followed by 5 mg/kg CQ base on the day of second and third injections and five days after the last placebo injection. Group B3 will undergo homologous CHMI with PfSPZ Challenge 10 weeks after the last immunization.
  Interventions: Biological: 0.9% Sodium Chloride (Placebo)

INTERVENTIONS:
Biological: PfSPZ Challenge — Aseptic, purified, vialed, cryopreserved, infectious P. falciparum sporozoites, strain NF54
  Arms: Stage A: Grp A1 - 3,200 PfSPZ Challenge; Stage A: Grp A2 - 12,800 PfSPZ Challenge; Stage A: Grp A3 - 51,200 PfSPZ Challenge; Stage B: Grp B1 - 51,200 PfSPZ Challenge; Stage B: Grp B2 - 51,200 PfSPZ Challenge; Stage B: Grp B3 - 51,200 PfSPZ Challenge
Biological: 0.9% Sodium Chloride (Placebo)
  Arms: Stage A: Grp A1 - 0.9% Sodium Chloride; Stage A: Grp A2 - 0.9% Sodium Chloride; Stage A: Grp A3 - 0.9% Sodium Chloride; Stage B: Group B1 - 0.9% Sodium Chloride; Stage B: Group B2 - 0.9% Sodium Chloride; Stage B: Group B3 - 0.9% Sodium Chloride

SUMMARY:
TÜCHMI-002 is a single center, randomized, placebo-controlled, double-blinded, PfSPZ Challenge dose finding trial with two chemoprophylactic regimens and subsequent controlled human malaria infection (CHMI).

DETAILED DESCRIPTION:
TÜCHMI-002 is a single center, randomized, placebo-controlled, double-blinded, PfSPZ Challenge dose finding trial with two chemoprophylactic regimens and subsequent controlled human malaria infection (CHMI), designed to establish a regimen of PfSPZ Challenge under chemoprophylaxis, with PfSPZ Challenge administered IV, that:

1. Is safe and well tolerated.
2. Provides consistent sterile protection against CHMI with homologous sporozoites in healthy adult subjects.
3. Is a practical regimen for PfSPZ Challenge chemoprophylaxis.

Volunteers will receive three immunizing PfSPZ Challenge IV injections 4 weeks apart under oral chemoprophylaxis. The trial is sequential and has two stages:

A) In the first stage, the PfSPZ Challenge dose is increased sequentially from 3,200 to 51,200 PfSPZ among the three groups. Controls for the three groups will receive 0.9% Sodium Chloride (NaCl) as placebo. All volunteers will receive a standard chemoprophylactic regimen of chloroquine (CQ) for 10 weeks. Briefly, 10 mg/kg CQ base will be given as loading dose followed by weekly doses of 5 mg/kg CQ base. Homologous CHMI is done with 3,200 PfSPZ Challenge IV eight weeks after the last immunizing PfSPZ Challenge injection.

B) In Stage B, accelerated regimens with CQ and CQ plus ER-AZ will be assessed. Initiation of Stage B of the trial is dependent upon demonstration of at least 75% (6 out of 8) protective efficacy against homologous CHMI in Stage A, no PfSPZ Challenge related SAEs and approval by the Safety Monitoring Committee (SMC). CHMI is done with 3,200 PfSPZ Challenge (NF54) IV ten weeks after the last immunization with PfSPZ Challenge under chemoprophylaxis. Injections are either done over 28 or 10 days, chemoprophylaxis is given for 5 weeks and 15 days, respectively. Control groups will receive 0.9% NaCl IV as placebo under the respective chemoprophylactic regimen.

Transition from Stage A to Stage B depends on a positive safety and efficacy review and approval by an independent SMC. Safety and efficacy data will also be submitted to the regulatory authorities (FDA in the U.S. and Paul-Ehrlich-Institute in Germany) as well as to the Ethics Committee. Sponsor, SMC and principal investigator will select PfSPZ dose after review of safety and efficacy data. In case of 100% efficacy of more than one dose regimen and comparable tolerability and safety, the higher PfSPZ dose will be used. Information about the selected dose together with the updated volunteer information document stating the dose will be submitted to the ethics committee for approval before initiation of Stage B. In case that PfSPZ Challenge related SAEs occur or efficacy of the best regimen is below 75% the study will not proceed to Stage B.

ELIGIBILITY:
Inclusion Criteria:

The volunteer must satisfy all the following criteria to be eligible for the study:

* Healthy adults aged 18 to 45 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the investigators to discuss the volunteer's medical history with their general practitioner ('Hausarzt') if required.
* Residence in Tübingen or surroundings for the period of the trial.
* Women only: Must agree to practice continuous effective contraception for the duration of the study (a method which results in a low failure rate; i.e. less than 1% per year).
* Agreement to refrain from blood donation during the course of the study and after the end of their involvement in the study according to the local and national blood banking eligibility criteria (currently four years in Germany).
* Written informed consent to receive PfSPZ Challenge for immunization and subsequently for CHMI.
* Reachable (24/7) by mobile phone during the immunization and CHMI period.
* Willingness to take CQ and ER-AZ during immunization and a curative antimalarial regimen following CHMI.
* Agreement to stay overnight for observation during the period of intensive follow-up post-challenge if required.
* Answer all questions on the informed consent quiz correctly.
* A body mass index <35.
* A hemoglobin concentration ≥12 g/dl for women and ≥13.5 g/dl for men.

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

* History of Pf malaria.
* Planned travel to malaria endemic areas.
* Use of systemic antibiotics with known antimalarial activity within 30 days of study enrollment (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones, or azithromycin).
* Receipt of an investigational product in the 30 days preceding enrollment, or planned receipt during the study period.
* Prior receipt of an investigational malaria vaccine.
* Immunization with more than 3 other vaccines within the past month.
* HIV infection.
* Any confirmed or suspected immunosuppressive or immunodeficient state, asplenia, recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* Presence of sickle cell anemia, sickle cell trait, thalassemia or thalassemia trait, glucose-6-phosphate dehydrogenase deficiency.
* Pregnancy, lactation or intention to become pregnant during the study.
* A history of allergic disease or reactions likely to be exacerbated by malaria.
* Contraindications to the use of the following antimalarial medications: atovaquone/proguanil, artemether-lumefantrine, mefloquine, azithromycin and chloroquine.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study (including but not restricted to organic, including symptomatic, mental disorders [ICD-10 code: F00-F09], schizophrenia, schizotypal and delusional disorders [F20-F29], mood (affective) disorders [F30-F39], mental retardation [F70-F79], Disorders of psychological development [F80-F89] or any other psychiatric condition that required hospitalization or psychiatric treatment over an extended period).
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 60 g (men) or 40 g (women) per day or a carbohydrate deficient transferrin (CDT) level ≥2.5%.
* Suspected or known injecting drug abuse in the 5 years preceding enrollment.
* Positive for hepatitis B surface antigen (HBs-antigen).
* Seropositive for hepatitis C virus (antibodies to HCV).
* Falling in moderate risk or higher categories for fatal or non-fatal cardiovascular event within 5 years (>10%) determined by non-invasive criteria for cardiac risk.
* Abnormal electrocardiogram on screening: pathologic Q wave and significant ST-T wave changes, left ventricular hypertrophy, non-sinus rhythm except isolated premature atrial contractions, right of left bundle branch block, advanced A-V heart block (secondary or tertiary).
* A QT/QTc interval >450 ms.
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or hematology blood tests, urine analysis or clinical examination.
* Retinal abnormalities.
* History of seizure.
* Any other significant disease, disorder or finding which, in the opinion of the investigator, may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

In case of inconclusive results of laboratory tests or other diagnostic procedures, test will be repeated. If doubts about the results persist, volunteers will be considered ineligible.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Proportion of volunteers who become parasitemic, detected by thick blood film microscopy, within 21 days following CHMI after immunization using PfSPZ Challenge or placebo under chemoprophylaxis [PfSPZ Challenge Vaccine (PfSPZ-CVac) approach]. | Within 21 days following CHMI
Occurrence of related Grade 3 adverse events (AEs) and SAEs from time of first administration of an immunizing regimen (chemoprophylactic antimalarial and PfSPZ Challenge) until the end of the study. | 19 months

SECONDARY OUTCOMES:
Time to microscopically detectable parasitemia (pre-patent period) in volunteers who become parasitemic within 21 days following CHMI after immunization using PfSPZ Challenge or placebo and an antimalarial. | Within 21 days following CHMI
Occurrence of any related AE from time of first administration of an immunizing regimen (chemoprophylactic antimalarial and PfSPZ Challenge) until the end of the study. | 19 months

OTHER OUTCOMES:
Proportion of participants who develop low-grade parasitemia, detected by quantitative polymerase chain reaction (qPCR), within 21 days following immunization with PfSPZ Challenge. | Within 21 days following CHMI
Occurrence of any (related and unrelated) AE from time of first administration of an antimalarial and PfSPZ Challenge until the end of the study. | 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Mordmüller, MD, Principal Investigator — Institute of Tropical Medicine, University of Tuebingen
Locations (1):
- Institute of Tropical Medicine, University of Tuebingen, Wilhelmstr. 27, Tübingen, Germany

REFERENCES:
- [Result] Mordmuller B, Surat G, Lagler H, Chakravarty S, Ishizuka AS, Lalremruata A, Gmeiner M, Campo JJ, Esen M, Ruben AJ, Held J, Calle CL, Mengue JB, Gebru T, Ibanez J, Sulyok M, James ER, Billingsley PF, Natasha KC, Manoj A, Murshedkar T, Gunasekera A, Eappen AG, Li T, Stafford RE, Li M, Felgner PL, Seder RA, Richie TL, Sim BK, Hoffman SL, Kremsner PG. Sterile protection against human malaria by chemoattenuated PfSPZ vaccine. Nature. 2017 Feb 23;542(7642):445-449. doi: 10.1038/nature21060. Epub 2017 Feb 15. PMID 28199305
- [Derived] Requena P, Gomez-Perez GP, McCall MBB, Barrios D, Aguilar R, Fernandez-Morata J, Vidal M, Campo JJ, Sanchez C, Yazdabankhsh M, Sim BKL, Hoffman SL, Kremsner P, Lell B, Mordmuller B, Dobano C, Moncunill G. Effect of controlled human Plasmodium falciparum infection on B cell subsets in individuals with different levels of malaria immunity. Med Microbiol Immunol. 2025 Sep 27;214(1):47. doi: 10.1007/s00430-025-00847-x. PMID 41014333